CLINICAL TRIAL: NCT01333436
Title: A Multicenter, Cross-sectional Study to Evaluate Plasma ApoB-48 Concentration Among Korean Diabetic Patients (With Normal to Moderately High LDL-C Levels)
Brief Title: A Study to Evaluate Fasting/Postprandial Serum Apolipoprotein B-48 (ApoB-48) Levels in Diabetic Participants With Normal to Moderately High Low Density Lipoprotein-C (LDL-C) Levels (MK-0653A-259 AM1)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 0653A-259
Record Dates: First submitted 2011-03-24; First posted 2011-04-12 (Estimated); Results first posted 2013-04-09 (Estimated); Last update posted 2024-05-13 (Actual); Status verified 2022-02

CONDITIONS: Dyslipidemia; Hypercholesterolemia
MeSH Terms: conditions — Dyslipidemias; Hypercholesterolemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Diabetic participants (Experimental): Diabetic participants with normal to moderately high LDL-C
  Interventions: Other: Test Meal
- Nondiabetic participants (Experimental): Non-diabetic participants with normal to moderately high LDL-C
  Interventions: Other: Test Meal

INTERVENTIONS:
Other: Test Meal — During Visit 2, a test meal will be supplied by the Sponsor of approximately 944 kcal (57% fat, 31% carbohydrate, and 12% protein), and postprandial blood draws will be done at 1, 2, 3, 4, and 6 hours after the meal.

SUMMARY:
This study will evaluate whether fasting/postprandial serum ApoB-48 levels are increased in diabetic participants compared to nondiabetic participants with the same range of serum LDL-C levels, and whether ApoB-48 levels can be used, along with LDL-C levels, to identify potential cardiovascular disease risk.

ELIGIBILITY:
Inclusion criteria:

* Participant has an LDL-C ranging from ≥100 mg/dL to <160 mg/dL.
* Patient has a triglyceride (TG) level of ≤500 mg/dL.

Exclusion Criteria:

* Participant treated with a lipid-lowering agent in the 6 weeks prior to Visit 1 (screening period).
* Participant has active liver disease or persistent unexplained serum transaminase elevations (≥2 x the upper limit of normal [ULN])
* Participant has increased creatine kinase (CK) (≥2 x ULN).
* Participant has a history of type 1 diabetes mellitus, ketoacidosis, or gestational diabetes mellitus.
* Participant has a history of alcohol and/or drug abuse.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2011-07-20 (Actual); Primary Completion 2012-05-12 (Actual); Study Completion 2012-05-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- MSD Korea Ltd., Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Park CY, Park JY, Choi J, Kim DJ, Park KS, Yoon KH, Lee MK, Park SW. Increased postprandial apolipoprotein B-48 level after a test meal in diabetic patients: A multicenter, cross-sectional study. Metabolism. 2016 Jun;65(6):843-51. doi: 10.1016/j.metabol.2016.02.008. Epub 2016 Feb 23. PMID 27173463

RESULTS

PARTICIPANT FLOW:
Groups:
- Diabetic Participants: Diabetic participants with normal to moderately high low-density lipoprotein-cholesterol (LDL-C) administered a test meal by the Sponsor during Visit 2 consisting of approximately 944 kcal (57% fat, 31% carbohydrate, and 12% protein).
- Nondiabetic Participants: Non-diabetic participants with normal to moderately high LDL-C administered a test meal by the Sponsor during Visit 2 consisting of approximately 944 kcal (57% fat, 31% carbohydrate, and 12% protein).
Period: Overall Study
Arm/Group | Diabetic Participants | Nondiabetic Participants
Started | 43 | 50
Completed | 43 | 50
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Diabetic Participants: Diabetic participants with normal to moderately high low-density lipoprotein-cholesterol (LDL-C) administered a test meal by the Sponsor during Visit 2 consisting of approximately 944 kcal (57% fat, 31% carbohydrate, and 12% protein.
- Nondiabetic Participants: Non-diabetic participants with normal to moderately high LDL-C administered a test meal by the Sponsor during Visit 2 consisting of approximately 944 kcal ( 57% fat, 31% carbohydrate, and 12% protein).
- Total: Total of all reporting groups
Arm/Group | Diabetic Participants | Nondiabetic Participants | Total
Number analyzed (Participants) | 43 | 50 | 93
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.0 (11.5) | 46.0 (13.6) | 49.7 (13.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 24 | 45
  Male | 22 | 26 | 48

OUTCOME MEASURES:

1. Primary Outcome: Postprandial Incremental Area Under the Curve From 0-6 Hours (iAUC)[0-6] of Apolipoprotein B-48 (ApoB-48)
Description: ApoB-48 levels were measured at 1, 2, 3, 4, and 6 hours after the administration of the test meal.
Time Frame: up to 6 hours after Test Meal
Population: Full-Analysis-Set (FAS) population defined as all participants who had valid postprandial ApoB-48 measurements for all specified time points to calculate iAUC.
Measure: Mean (Standard Deviation); unit: μg/mL x h
Arm/Group | Diabetic Participants | Nondiabetic Participants
Number analyzed (Participants) | 42 | 46
μg/mL x h | 63.4 (42.4) | 41.7 (30.9)
Statistical Analysis 1: Comparison: Diabetic Participants vs Nondiabetic Participants; Test type: Superiority or Other; p = 0.0078, t-test, 2 sided; Mean Difference (Final Values) = 21.8, Standard Deviation 36.8

2. Secondary Outcome: Postprandial Mean ApoB-48 Peak Levels
Description: ApoB-48 levels measured at 1, 2, 3, 4, and 6 hours after the administration of test meal. Peak was the highest ApoB-48 level recorded during this timeframe.
Time Frame: up to 6 hours after Test Meal
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | Diabetic Participants | Nondiabetic Participants
Number analyzed (Participants) | 42 | 46
μg/mL | 24.8 (15.7) | 19.3 (11.9)
Statistical Analysis 1: Comparison: Diabetic Participants vs Nondiabetic Participants; Test type: Superiority or Other; p = 0.0675, t-test, 2 sided; Mean Difference (Net) = 5.5, Standard Deviation 13.9

3. Secondary Outcome: Fasting ApoB-48 Levels
Description: ApoB-48 levels measured after at least a 12-hour fast and prior to administration of test meal (Hour 0).
Time Frame: Baseline (Hour 0)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | Diabetic Participants | Nondiabetic Participants
Number analyzed (Participants) | 42 | 46
μg/mL | 5.9 (3.5) | 7.3 (5.8)
Statistical Analysis 1: Comparison: Diabetic Participants vs Nondiabetic Participants; Test type: Superiority or Other; p = 0.1798, t-test, 2 sided; Mean Difference (Net) = -1.4, Standard Deviation 4.8

ADVERSE EVENTS:
Arm/Group | Diabetic Participants | Nondiabetic Participants
Serious Adverse Events (participants affected / at risk) | 0/43 | 0/50
Other Adverse Events (participants affected / at risk) | 0/43 | 0/50

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Subsequent to the multicenter publication, or 24 months after completion of the study, whichever comes first, an investigator and/or his/her colleagues may publish the results for their study site independently. The SPONSOR must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation.